CLINICAL TRIAL: NCT00003003
Title: A Pilot Clinical Trial of Mitomycin C Modulation of Multidrug Resistance Proteins and a Phase I Evaluation of Mitomycin C and Mitoxantrone in Patients With Acute Myelogenous Leukemia
Brief Title: Mitomycin and Mitoxantrone in Treating Patients With Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher H. Lowrey, Hematology Oncologist, Dartmouth-Hitchcock Medical Center
Purpose: Treatment
Other Study IDs: CDR0000065565; P30CA023108 (NIH); DMS-9614; NCI-V97-1260
Record Dates: First submitted 1999-11-01; First posted 2004-08-12 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2000-06

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — sargramostim; Mitomycin; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: sargramostim
Drug: mitomycin C
Drug: mitoxantrone hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Some cancers become resistant to chemotherapy drugs. Combining mitomycin with a chemotherapy drug may reduce resistance to the drug and allow the cancer cells to be killed.

PURPOSE: Phase I trial to study the effectiveness of mitomycin and mitoxantrone in treating patients with acute myelogenous leukemia and to determine whether mitomycin can reduce the cancer's resistance to chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether a single mitomycin C treatment will suppress expression of one or more proteins associated with the multidrug resistance phenotype in leukemia cells of patients with refractory acute myelogenous leukemia. II. Determine the maximum tolerated dose of a combination of mitomycin C followed 72 hours later by a single dose of mitoxantrone in patients with acute myelogenous leukemia with GM-CSF support. III. Determine the toxicity profile and pharmokinetics for these combinations of mitomycin C and mitoxantrone. IV. Determine the ability of this regimen to induce complete response in patients with primary resistant or refractory acute myelogenous leukemia.

OUTLINE: Patients receive mitomycin C by IV bolus on day 1 of treatment. Patients receive mitoxantrone beginning on day 4. One patient each is entered at the first and second dose levels. Dose escalation of mitoxantrone continues in the absence of toxicity. If the patient experiences toxicity at level 1 or 2, then 2 additional patients are entered at that tier. Three patients are entered at all subsequent tiers. At these tiers, if no toxicity is observed, escalation continues. If 1 of the 3 patients experiences toxicity, an additional 3 patients are enrolled at the same dose. If none of these additional patients experiences toxicity, escalation continues; however, if 1 patient has toxicity, the trial is stopped. If 2 or more have toxicities, the dose is de-escalated. If 2 or more of the original 3 patients have toxicities, the dose is de-escalated. On day 15, patients are treated with sargramostim (GM-CSF) intravenously over 4 hours if the bone marrow is free of residual leukemia; GM-CSF treatment continues until the ANC is greater than 1,500/mm3 for 3 consecutive days.

PROJECTED ACCRUAL: For the pilot study of mitomycin C modulation of multidrug resistance proteins, 12 patients will be accrued. For the phase I study of mitomycin C and mitoxantrone, at least 17 patients will be entered.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Acute myelogenous leukemia, either de novo or secondary (evolving from myelodysplastic syndrome, myeloproliferative syndrome, or previous treatment for malignancies other than leukemia) OR Refractory anemia with excess blasts in transformation Patient is at least 60 years old and at least one of the following is true: Failed one induction attempt or First or greater relapse OR Patient is 18-59 years old without an acceptable allogeneic donor and no autologous marrow for transplant and at least one of the following is true: Failed 2 separate induction attempts, or Second or greater relapse, or Resistant relapse, or Relapsed post transplant Prior treatment with anthracyclines or mitoxantrone required Cumulative daunorubicin dose less than 400/m2 required

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70%-100% (50% if hospitalized) Hematopoietic: Not specified Hepatic: Total direct bilirubin no greater than 2.0 mg/dL SGOT and SGPT no greater than 3 x normal Alkaline phosphatase no greater than 3 x normal No active hepatitis Renal: Not specified Cardiovascular: No myocardial infarction within last 6 months No congestive heart failure Ejection fraction greater than 50% (measured by MUGA or 2-D Echo) Pulmonary: No severe chronic obstructive pulmonary disease Other: No active infection or antimicrobiologically stabilized infection Not pregnant

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 1996-09; Primary Completion 2000-08 (Actual); Study Completion 2000-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher H. Lowrey, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Norris Cotton Cancer Center, Lebanon, New Hampshire, United States